CLINICAL TRIAL: NCT02101541
Title: Focal Impulse and Rotor Modulation (FIRM) as a Stand-alone Procedure in the Treatment of Atrial Fibrillation
Brief Title: FIRM as a Stand-alone Procedure in the Treatment of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Rolf Franck Berntsen, M.D, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/627
Record Dates: First submitted 2014-02-28; First posted 2014-04-02 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Arrhythmias, Cardiac; Heart diseases; Cardiovascular diseases; Pathological processes
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FIRM ablation (Experimental): The first part of this within-patient trial investigate the efficacy of focal impulse and rotor modulation in 20 patients with paroxysmal atrial fibrillation, evaluated by continuous pre- and post-procedural heart rhythm monitoring.
  The second part consists of 20 patients with persistent or longstanding persistent atrial fibrillation following the same scheme.
  Interventions: Procedure: FIRM ablation

INTERVENTIONS:
Procedure: FIRM ablation — Radiofrequency catheter ablation of atrial fibrillation driving sources detected by sequential bi-atrial panoramic contact mapping.
  Other Names: Atrial fibrillation; Rotors; Mapping; Radiofrequency ablation

SUMMARY:
The FIRM Study Oslo will in two sequential within-patient trials investigate the efficacy of focal impulse and rotor modulation (FIRM) as a stand-alone procedure in the treatment of paroxysmal and persistent atrial fibrillation, evaluated by continuous pre- and post-procedural heart rhythm monitoring.

DETAILED DESCRIPTION:
After a pilot/implementation study consisting of 10 patients with paroxysmal atrial fibrillation (AF); 20 patients with paroxysmal AF will be included in a within-patient trial. This study will be followed by a similar comparison in 20 patients with persistent or longstanding persistent AF.

The AF driving sources will be visualized by a novel sequential bi-atrial panoramic contact mapping technique. Unipolar signals will be recorded by a 64-polar basket catheter (FIRMap®, Topera. Inc.), then processed and the activation patterns visualized (RhythmView® 3D Electrophysiologic Mapping System, Topera, Inc.).

Focal impulse and rotor modulation (FIRM) will then be performed with standard irrigated radio frequency catheter ablation until rotor or focal impulse elimination is confirmed by repeat FIRM mapping.

Treatment efficacy will be assessed with continuous heart rhythm monitors (Reveal XT®, Medtronic, Minneapolis, USA) implanted 3 months prior to ablation, and freedom from AF defined as AF burden <1% at follow-up at 12, 24 and 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation despite of at least one Class I or Class III antiarrhythmic drug and/or previous conventional ablation (pulmonary vein isolation).
* At least one episode of paroxysmal atrial fibrillation should be documented by rhythm strip, ECG or implanted monitor during the last 6 months prior to ablation.

Exclusion Criteria:

* Significant structural heart disease (including symptomatic coronary heart disease; prosthetic mitral or tricuspid valve; congenital heart disease where abnormality or its correction prohibits or increases the risk of ablation).
* Intracardiac thrombus, tumor or dense contrast on TEE.
* Contraindication to anticoagulant therapy (heparin, warfarin, dabigatran and rivaroxaban).
* Anaphylactic allergy to contrast media.
* Poor general health resulting from other disease.
* Inability or refusal to provide written informed consent for the study.

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Single procedure freedom from atrial fibrillation (AF) at 12 months. | 12 months.
  Freedom from AF defined as <1% AF burden as detected by the implanted heart rhythm monitor.

SECONDARY OUTCOMES:
Single procedure freedom from atrial fibrillation (AF) at 24 months. | 24 months.
  Freedom from AF defined as <1% AF burden as detected by the implanted heart rhythm monitor.
Single procedure freedom from atrial fibrillation (AF) at 30 months. | 30 months.
  Freedom from AF defined as <1% AF burden as detected by the implanted heart rhythm monitor.

OTHER OUTCOMES:
Cumulative freedom from atrial fibrillation (AF) (multi-procedure). | 30 months.
  Cumulative freedom from AF (multi-procedure) measured from final study.
Major procedure related events. | 0 to 12 months.
  Cardiac tamponade/perforation; stroke; transient ischemic attack; bleeding; vascular access complications; injury to the esophagus/phrenic or vagal nerve etc.
Number of rotors identified and percentage eliminated on remap. | Procedural.
  Number of rotors identified and percentage eliminated on remap will be evaluated during the procedure.
Quality of life (QOL). | 12 months.
  QOL will be evaluated by the SF-36 health survey (Norwegian version) pre- and 12 months post ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Franck Berntsen, MD, PhD, Principal Investigator — Dept. of Cardiology, Rikshospitalet - Oslo University Hospital
Locations (1):
- Dept. of Cardiology, Rikshospitalet - Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No